CLINICAL TRIAL: NCT03214276
Title: Effects of Acute Specific Grape and Apple Polyphenols Supplementation on Cycling Endurance Performance
Brief Title: Effects of Polyphenols Supplementation on Cycling Endurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Burgundy (Other)
Responsible Party: Principal Investigator, Nicolas Babault, Principal investigator, University of Burgundy
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CEN1143
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: polyphenols; cycling; endurance; aerobic; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyphenols (Active Comparator): The preceding night and one hour before the endurance test, participants were asked to absorb two capsules of 250 mg of polyphenols (Vinitrox™)
  Interventions: Dietary Supplement: Vinitrox polyphenols
- placebo (Placebo Comparator): The preceding night and one hour before the endurance test, participants were asked to absorb two capsules of placebo (similar appearance and flavour than active comparator).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vinitrox polyphenols — Vinitrox™ (Nexira - France) is a combination of specific profile polyphenols from grape and apple. The main polyphenol classes are proanthocyanidins (as catechins, B2 dimer), phenolic acids (as chlorogenic acids, gallic acids) and anthocyanins (as malvidin-3-glucoside). It was administrated the night and the morning before the endurance test (oral administration)
  Arms: Polyphenols
Dietary Supplement: Placebo — Made with maltodextrin. It was administrated the night and the morning before the endurance test (oral administration).
  Arms: placebo

SUMMARY:
Endurance performance during high intensive exercises is mainly determined by the capacity of the aerobic metabolism. It generally induces muscle fatigue defined as the reversible decline in skeletal muscle contractile performance. Fatigue is multifactorial and is often associated with many physiological parameters including reduced neural input and disruptive metabolic changes in skeletal muscles such as lactic acidosis and the production of oxidative free radicals. Moreover, it could lead to oxidative stress as a result of an imbalance between reactive oxygen species (ROS) production and intrinsic antioxidant defense.

To alleviate oxidative stress, some ergogenic strategies have been tested. Numerous studies have reported that different types of supplementation such as selenium, vitamin E, vitamin C or polyphenols were of interest to protect against these mechanisms. Indeed, although some studies demonstrated no or harmful effects, most studies observed positive effects of antioxidants on oxidative stress or performance. More particularly, polyphenols, have great antioxidant capabilities and protective effects and it increases the synthesis and bioavailability of nitric oxide (NO)which is well known to be the most important mediator of vasodilation. To date, most of the studies exploring the effects of polyphenols on exercise investigated several days or weeks of supplementations on vascular, blood parameters (blood pressure, NO concentration, oxidative stress markers) or endurance performance. Conflicting results are often obtained. Only few studies investigated the effects of a single intake on immediate performance and recovery capacity. Therefore, the present work aimed to study the effects of an acute intake of a specific profile polyphenols from grape and apple on physical performances. More specifically, performance, in the present study, referred to high intensity cycling exercise until exhaustion revealing the capacity to maintain a constant strong effort hereafter named endurance. The hypothesis was that an acute of polyphenols would increase the time to exhaustion during a high intensity cycling exercise.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index lower than 27 and waist size lower than 94 cm
* physical activity higher than 2 hours a week
* written informed consent

Exclusion Criteria:

* more than 6 hours training a week, regularly trained in aerobic activities
* asthmatic, smokers or under medicinal drugs
* dietary supplement, sports drink, special dietary food or functional food, of any kind, liable or presented as liable to enhance physical performances

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2012-07-01 (Actual)

PRIMARY OUTCOMES:
Time to exhaustion | The total duration of the aerobic exercise (during the cycling aerobic exercise)
  Maximal duration during a cycling aerobic exercise (70% of maximal aerobic power)

SECONDARY OUTCOMES:
Heart rate | Immediately before the endurance test, immediately after the endurance test and continuously recorded during three minutes during the recovery to determine half-recovery time
  Heart rate using a polar belt
Gaz exchange | Immediately before the endurance test, immediately after the endurance test and continuously recorded during three minutes during the recovery to determine half-recovery time
  oxygen intake using a portable gaz exchange analyzer
blood pressure | Immediately before the endurance test, immediately after the endurance test
  blood pressure measured at the arm
Pain sensation | Immediately after the endurance exercise and 48 hours after the endurance test
  Pain sensation using a visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Babault, PhD, Principal Investigator — University of Burgundy

IPD SHARING:
Plan to Share IPD: No